CLINICAL TRIAL: NCT04560556
Title: Linking Persons With HIV, Discharged From Jail, With Community Care: a Direct Comparison of the Costs and Effects of Three HIV Management Strategies in the District of Columbia Department of Corrections
Brief Title: Linking Persons With HIV, Discharged From Jail, With Community Care
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Anne C Spaulding, Associate Professor, Emory University
Other Study IDs: IRB00115929
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Correctional settings; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- POC Testing Alone: POC HIV testing (the current standard of care) will be conducted for persons entering jail during the first two-month period.
  Interventions: Diagnostic Test: Point-of-Care (POC) Rapid HIV Test
- POC and 4th Generation Testing: POC plus 4th Generation HIV Testing will be conducted for persons entering jail during the second two-month period.
  Interventions: Diagnostic Test: Point-of-Care (POC) Rapid HIV Test; Diagnostic Test: Fourth Generation Antigen/antibody (Ag/Ab) HIV Test
- 4th Generation Testing Alone: 4th Generation HIV Testing will be conducted for persons entering jail during the third two-month period.
  Interventions: Diagnostic Test: Fourth Generation Antigen/antibody (Ag/Ab) HIV Test

INTERVENTIONS:
Diagnostic Test: Point-of-Care (POC) Rapid HIV Test — Point-of-care (POC) rapid HIV testing provides results within minutes, however, it cannot reliably detect new infections. It can take up to 90 days after exposure for HIV infections to be diagnosed with POC rapid testing.
  Groups: POC Testing Alone; POC and 4th Generation Testing
Diagnostic Test: Fourth Generation Antigen/antibody (Ag/Ab) HIV Test — Fourth generation laboratory-based antigen/antibody (Ag/Ab) HIV testing can detect acute HIV infections (as early as 18 days after exposure), but it takes several hours to process.
  Groups: 4th Generation Testing Alone; POC and 4th Generation Testing

SUMMARY:
This is a prospective cohort study of outcomes of individuals who entered jail during a period during which one of three serial HIV testing strategies is implemented. This study involves two sub-studies. One sub-study will examine referrals to HIV prevention programs for persons testing negative for HIV while in jail. The second sub-study will monitor antiviral use among those testing positive for HIV.

DETAILED DESCRIPTION:
Incarcerated Americans on any given day represent one in 40 (2.5%) Persons Living with HIV (PLWH) in this country, but those ever incarcerated over the course of a year represent 17% of the US epidemic. PLWH are a diverse group in terms of awareness and management of their disease. A portion may be aware of their HIV status and on treatment. This subgroup is at risk of disruption in care if incarcerated. Others may be aware of their status, but untreated, while still others may be unaware of their HIV status. The latter group is of particular importance in terms of the HIV epidemic in criminal justice settings, as a recent meta-analysis indicated that up to 15% of individuals entering jail have undiagnosed infections.

Good management of PLWH during a period of incarceration is critical. Ensuring that care relationships are maintained or newly established will improve health outcomes among PLWH and reduce the risk of transmission once they are discharged. As the median length of stay in jail is short (median < 7 days), rapid HIV testing is critical. Maximizing the yield and speed of HIV testing in a jail environment has the potential to promote rapid entry into care, or rapid re-engagement if persons have fallen out of care. For those testing negative, it can hasten the referral to Pre-Exposure Prophylaxis (PrEP) services.

How correctional facilities offer HIV testing and begin treatment affects long-term outcomes. Because of the rapid churn of jail, point-of-care (POC) rapid testing may lead to a higher percentage of patients receiving test results before leaving jail, compared to conventional assays. Fourth generation laboratory-based antigen/antibody (Ag/Ab) testing can diagnosis more persons with acute HIV infection, who may be in the window period before the POC test turns positive, but has a several hour test turn-around time, and those tested may leave jail before receiving their result. Using both tests for every entrant would permit the jail to experience the benefit of both methods but at greater expense. Collaborating with Washington, DC's city jail, known as DC Department of Corrections (DC DOC), and Unity Healthcare, the network of Federally Qualified Health Centers in Washington DC, which also provides care within the DC DOC, this study has a unique opportunity to measure rapidity of testing, linkage to and commencement of care, and achievement of viral suppression, along with costs of HIV identification.

This study uses a unique, time-sensitive opportunity to compare three separate strategies of universal HIV screening and treating. The strategies of POC testing, 4th generation laboratory-based Ag/Ab testing, and a combination of the two tests will be compared in the DC jail. A rigorous assessment of the three strategies in terms of their feasibility, process measures, and cost-effectiveness on an institutional level will help to guide implementation decisions in jails across the US.

One sub-study will assess the number of persons testing negative who are referred to prevention programs after leaving the jail. A second sub-study will examine antiviral use after jail release, among PLWH.

ELIGIBILITY:
Inclusion Criteria for Those Testing Negative for HIV:

* Able to understand and speak English
* Confirmed HIV negative status
* Planning to stay in the metropolitan DC area upon jail release
* Candidate for PrEP using attached screening instrument and interested in taking it

Inclusion Criteria for Those Testing Positive for HIV:

* Able to understand and speak English
* Confirmed HIV positive status
* Planning to stay in the metropolitan DC area upon jail release

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from the study population of NCT04296331, comprised of individuals admitted to D.C. Central Detention Facility (DC DOC) between October 2019 and April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Number of Entrants Tested | Up to 24 hours
  The number of entrants receiving an HIV test within 24 hours of intake will be examined.
Percentage of PLWH Identified in First 24 Hours | Up to 24 hours
  The percentage of PLWH identified within the first 24 hours of admission, among all PLWH who enter, will be examined.
Number of New HIV Diagnosed Prior to Discharge | Up to Jail Discharge
  The number of persons with a new diagnosis of HIV who receive test results before discharge will be examined.
Number of Entrants with Acute HIV Infection Identified | Up to 5 days
  The number of entrants identified having an acute HIV infection will be examined.

SECONDARY OUTCOMES:
Time Until Receipt of Positive Test Result | Up to 5 days
  The time (in hours) from the positive test result in persons not previously diagnosed and receipt of test report.
Time Until Receipt of Antiviral Dose | Up to Jail Discharge
  The time (in days) from entry until receipt of first dose of antiviral in the jail, for PLWH.
Time Until Viral Suppression | 6 months after positive HIV intake test
  For all PLWH, the time (in days) from entry to achieving viral suppression, if not suppressed at baseline.
Time Until Meeting with Discharge Planner | Up to Jail Discharge
  For all PLWH, the time (in days) from intake to meeting the discharge planner.
Number of Participants Taking PrEP | 2 months after jail release, 6 months after jail release
  For those consenting to the first sub-study, the number of high-risk persons who test negative for HIV who successfully link to PrEP within 2 months of jail release and stay on PrEP for at least 6 months will be examined.
Number of PLWH who Attend Clinic Visits | 1 year
  For persons living with HIV who consent to the second sub-study, the percentage of persons previously and newly diagnosed who make clinic visits at least once every 6 months will be examined.
Number of PLWH with Viral Suppression | 6 months
  For persons living with HIV who consent to the second sub-study, the percentage of persons previously and newly diagnosed who are virally suppressed 6 months after sub-study enrollment.
Cost of Each Testing Strategy | 6 months
  A cost-effectiveness analysis using the intermediate process measures will be conducted. Units of resource items, such as tests and staff time, will be multiplied by their unit costs to calculate total costs. Wage ranges provided by DOC and Unity Healthcare will be used to price staff time; market values will be used for all other items. Costs will then be summed by testing strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Spaulding, MD, MPH, Principal Investigator — Emory University
Locations (1):
- DC Department of Corrections, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified laboratory results, demographics, and survey questions may be made available to other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will available for sharing after publication of the main article from this study.
Access Criteria: Individual participant data will be available for sharing with fellow researchers who submit a proposal for secondary data analysis. Proposals should be sent to aspauld@emory.edu.